CLINICAL TRIAL: NCT02733484
Title: Probiotics Effect on Glucose and Lipid Metabolism and Gut Microbiota in Patients With Obesity: a Randomized, Double-blind Controlled Trial
Brief Title: Probiotics Effect on Glucose and Lipid Metabolism and Gut Microbiota in Patients With Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Huanlong Qin, Professor, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PTD02
Record Dates: First submitted 2016-04-05; First posted 2016-04-11 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Obesity
Keywords: Obesity,Probiotics,Treatment
MeSH Terms: conditions — Obesity | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotics (Experimental): the patients in this arm will receive probiotics with a dose for 2g/d for 3 months.
  Interventions: Dietary Supplement: Probiotics
- Placebo (Placebo Comparator): the patients in this arm will receive placebo with similar appearance of probiotics.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics — the patients in this arm will receive probiotics with a dose for 2g/d for 3 months.
  Arms: Probiotics
Dietary Supplement: Placebo — the patients in this arm will receive placebo intervention
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether the probiotics will be effective in the treatment of obesity

DETAILED DESCRIPTION:
This study aims to evaluate the effect of probiotics on the improvement of glucose and lipid metabolism, as well as the gut microbiota.Baseline, 1 month and 3 months data will be collected and put into analysis to provide some suggestions on the probiotics use in the clinical practice for obesity patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 15-60 years
2. BMI≥28.0kg/m2
3. Agree to cooperate in the trial
4. Provision of written informed consent

Exclusion Criteria:

1. With chronic gastrointestinal diseases, severe immune deficiency, lactose intolerance
2. Diabetes
3. Use antibiotics, bacteriostatic agents (eg berberine), lipid-lowering drugs, antacids, H2 Blockers, proton pump inhibitors, corticosteroids or sex hormones
4. Use any probiotics in the last 3 months
5. Allergic constitution
6. Participating in any other clinical trials
7. Was not able to insist until the end
8. Pregnant and lactating women

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
change from baseline in fasting blood-glucose at 1 month | 1 month
  change of the fasting blood-glucose will be calculated at 1 month in comparison with the baseline
change from baseline in fasting blood-glucose at 3 months | 3 months
  change of the fasting blood-glucose will be calculated at 3 months in comparison with the baseline
change from baseline in glycosylated hemoglobin change at 1 month | 1 month
  change of the glycosylated hemoglobin will be calculated at 1 month in comparison with the baseline
change from baseline in glycosylated hemoglobin change at 3 months | 3 months
  change of the glycosylated hemoglobin will be calculated at 3 months in comparison with the baseline

SECONDARY OUTCOMES:
change from baseline in gut microbiota at 1 month | 1 month
  study the microbiota change of stool samples at 1 month in comparison with the baseline
change from baseline in gut microbiota at 3 months | 3 months
  study the microbiota change of stool samples at 3 months in comparison with the baseline
change from baseline in triglyceride at 1 month | 1 month
change from baseline in triglyceride at 3 months | 3 months
change from baseline in cholesterol at 1 month | 1 month
change from baseline in cholesterol at 3 months | 3 months
change from baseline in high-density lipoprotein at 1 month | 1 month
change from baseline in high-density lipoprotein at 3 months | 3 months
change from baseline in low-density lipoprotein at 1 month | 1 month
change from baseline in low-density lipoprotein at 3 months | 3 months
change from baseline in glutamic oxalacetic transaminase at 1 month | 1 month
change from baseline in glutamic oxalacetic transaminase at 3 months | 3 months
change from baseline in alkaline transaminase at 1 month | 1 month
change from baseline in alkaline transaminase at 3 months | 3 months
change from baseline in alkaline phosphatase at 1 month | 1 month
change from baseline in alkaline phosphatase at 3 months | 3 months
change from baseline in superoxide dismutase at 1 month | 1 month
change from baseline in superoxide dismutase at 3 months | 3 months
change from baseline in C-reactive protein at 1 month | 1 month
change from baseline in C-reactive protein at 3 months | 3 months
change from baseline in uric acid at 1 month | 1 month
change from baseline in uric acid at 3 months | 3 months
change from baseline in tumor necrosis factor-a at 1 month | 1 month
change from baseline in tumor necrosis factor-a at 3 months | 3 months
change from baseline in interleukin-6 at 1 month | 1 month
change from baseline in interleukin-6 at 3 months | 3 months
change from baseline in interleukin-8 at 1 month | 1 month
change from baseline in interleukin-8 at 3 months | 3 months
change from baseline in fasting insulin at 1 month | 1 month
change from baseline in fasting insulin at 3 months | 3 months
change from baseline in c peptide at 1 month | 1 month
change from baseline in c peptide at 3 months | 3 months
change from baseline in visceral fat fraction at 1 month | 1 month
change from baseline in visceral fat fraction at 3 months | 3 months
change from baseline in body age at 1 month | 1 month
change from baseline in body age at 3 months | 3 months
change from baseline in percentage of body fat at 1 month | 1 month
change from baseline in percentage of body fat at 3 months | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Huanlong Qin, Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Shanghai 10th People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided